CLINICAL TRIAL: NCT05361746
Title: Clinical Performance of a New Dental Adhesive, 3M™ Scotchbond™ Universal Plus Adhesive, Compared to 3M™ Scotchbond™ Universal Adhesive When Used With 3M™ Filtek™ Universal Restorative to Restore Class V Non-carious Cervical Lesions
Brief Title: Scotchbond Universal Plus Compared to Scotchbond Universal With Filtek Universal Restorative to Restore Class V NCCLs
Acronym: SBU+ClassV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EM-11-050068
Record Dates: First submitted 2022-04-30; First posted 2022-05-05 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Class V Non-carious Cervical Dental Lesions
Keywords: composite resins; dental adhesives; noncarious lesions; abfraction lesions; bonding, dental; clinical study; Scotchbond Universal plus; Scotchbond Universal; Filtek; dental materials

STUDY DESIGN:
Intervention Model Description: Each subject will have either two restorations (two teeth) or four restorations (four teeth) performed at the beginning of the study, with each tooth restoration using only one type of adhesive. Study teeth will be paired according to lesion depth and randomized to treatment in a 1:1 ratio with at least half of the teeth (ie, 1 tooth for Subjects with 2 eligible teeth or 2 teeth for Subjects with 4 eligible teeth) randomized to undergo restoration(s) using Scotchbond Universal Plus Adhesive (SBU+ Treatment group) and the other half of the teeth undergoing restoration(s) using Scotchbond Universal Adhesive (SBU Control group).
Who Masked: Outcomes Assessor
Masking Description: All assessments will be performed by two dental examiners that are independent of the dentist that placed the restorations and are blinded to the treatment arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SBU+ Treatment Group (Experimental): Either 1 tooth (for Subjects with 2 eligible teeth) or 2 teeth (for Subjects with 4 eligible teeth) with Class-V NCCLs will undergo restoration(s) using Scotchbond Universal Plus (SBU+) Adhesive .
  Interventions: Device: Scotchbond Universal Plus Adhesive
- SBU Control Group (Active Comparator): Either 1 tooth (for Subjects with 2 eligible teeth) or 2 teeth (for Subjects with 4 eligible teeth) with Class-V NCCLs will undergo restoration(s) using the predicate device, Scotchbond Universal (SBU) Adhesive.
  Interventions: Device: Scotchbond Universal Adhesive

INTERVENTIONS:
Device: Scotchbond Universal Plus Adhesive — Eligible teeth with Class-V NCCLs randomized to the SBU+ treatment group will undergo restoration(s) using Scotchbond Universal Plus (SBU+) Adhesive using total-etch mode and Filtek Universal Restorative material.
  Arms: SBU+ Treatment Group
Device: Scotchbond Universal Adhesive — Eligible teeth with Class-V NCCLs randomized to the SBU Control group will undergo restoration(s) using Scotchbond Universal Plus (SBU) Adhesive using total-etch mode and Filtek Universal Restorative material.
  Arms: SBU Control Group

SUMMARY:
This is a prospective, controlled, within-subject, randomized, single-center study comparing Scotchbond Universal Plus and Scotchbond Universal adhesives when used with Filtek restorative. The study will enroll a minimum of 46 Subjects with Class-V non-carious cervical lesion (NCCL) on a minimum of two teeth.

DETAILED DESCRIPTION:
This is a prospective, controlled, within-subject, randomized, single-center study that will enroll Subjects scheduled to undergo Class-V NCCL restorations on 2 or 4 teeth treated in pairs according to lesion depth. The study will enroll a minimum of 46 Subjects from a single site located in Birmingham, AL, USA. Each study tooth will be restored using only one type of adhesive, either SBU+ or SBU, and Filtek restorative. Any teeth needing treatment that are not included in the study will be treated by the dentist using the standard of care.

Subjects will be seen during screening (≤21 days before the restoration procedure), on the day of the restoration procedure, 7 days (± 3 days) after restoration (remote visit for subject self-assessment of baseline hypersensitivity), and follow-up visits at 6 months (± 14 days), 1 year (± 30 days), and 2 years (± 45 days) after restorations. Study teeth will be assessed for selected endpoints based partly on FDI World Dental Federation criteria. Subjects may participate in additional unscheduled visits as required during the study if evaluation of any study tooth is required outside of the scheduled study visits. The entire duration of the study is expected to last approximately 3 years, with individual Subject participation expected to last up to 2 years (± 45 days).

To help minimize or avoid bias in the study, randomization of study teeth will occur after teeth preparation but before the initial application of any adhesive. All assessments will be performed by 2 dental examiners that are independent of the dentist that placed the restorations and are blinded to the treatment arms. All examiners will be trained and calibrated for the scoring criteria before any Subject assessment occurs, and examiners will be retrained and recalibrated if any new evaluator is added to the list of assessors. After the second examiner has completed their assessments, the examiners will compare their evaluations and a consensus will be reached for each of the scoring criteria at each visit before the Subject leaves the visit. The consensus assessments will be entered into the Case Report Form (CRF).

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included that meet the following criteria:

1. Subject is at least 18 years of age at the time of consent
2. Subject is able to provide their own informed consent
3. Subject has a minimum of two teeth that:

   * have non-carious Class V lesions that are at least 1.5 mm deep
   * are not devitalized
   * have not undergone root canal treatment
4. Subject has an Approximal Plaque Index score ≤ 40% as assessed via explorer and without the use of plaque-disclosing agents
5. Subject is able and willing to return for all scheduled study visits
6. Subject meets the Level-I or Level-II classification criteria of the American Society of Anesthesiologists (ASA) Physical Status Classification System For Dental Patient Care

Exclusion Criteria:

Subjects may not be included that meet any of the following criteria:

1. Subject has any of the following:

   * rampant caries
   * chronic periodontitis
   * salivary gland dysfunction
2. Subject is unable, for any reason, to tolerate the procedure time required to place the restorations
3. Subject has unacceptable oral hygiene (eg, chronic moderate to heavy plaque accumulation along the gumline)
4. Subject has known sensitivity to the study product components (ie, acrylate)
5. Subject is planned to be enrolled in another investigational trial that requires additional interventions at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Restoration Retention | 24 months
  proportion of Subjects with partial or complete loss of the restoration materials
Marginal Adaptation | 24 months
  Marginal adaptation / marginal integrity of restorations scored on scale of 1-5

SECONDARY OUTCOMES:
Restoration Retention | baseline, 6 months, 12 months
  proportion of Subjects with partial or complete loss of the restoration material
Marginal Adaptation | baseline, 6 months, 12 months
  Marginal adaptation / marginal integrity of restorations scored on scale of 1-5
Fracture of Restorative Material | baseline, 6 months, 12 months, 24 months
  Fractures on study teeth scored on a scale of 1-4
Secondary Caries | baseline, 6 months, 12 months, 24 months
  Incidence of secondary caries of study teeth scored on scale 1-5

OTHER OUTCOMES:
Surface staining | baseline, 6 months, 12 months, 24 months
  Surface staining of study teeth scored on a scale of 1-5
Marginal staining | baseline, 6 months, 12 months, 24 months
  Marginal staining of study teeth scored on a scale of 1-5
Color match | baseline, 6 months, 12 months, 24 months
  Color match and translucency of study teeth on a scale of 1-5
Polish retention | baseline, 6 months, 12 months, 24 months
  Polish retention (surface gloss / luster and roughness) scored on a scale of 1-7
Post-operative hypersensitivity and tooth vitality | 6 months, 12 months, 24 months
  Post-operative hypersensitivity and tooth vitality upon exposure of the study teeth to a cold cotton pellet scored on a scale of 1-5
Time to restoration failure | 24 months
  Restoration retention survival time defined as the time between the restoration date and the first report of the presence of restoration failure
Patient satisfaction | baseline, 6 months, 12 months, 24 months
  Survey of patient satisfaction with aesthetics and function of tooth restorations
Incidence of adverse events | 24 months
  Adverse device effects collected from time of restoration through 24-month follow-up visit
Baseline post-operative hypersensitivity (subject self-assessment) | 7 days
  Post-operative hypersensitivity assessed at baseline by the subject on a scale of 1-3

CONTACTS AND LOCATIONS:
Overall Officials: John Burgess, DDS, MS, Principal Investigator — Louisiana State University HSC Health, School of Dentistry
Locations (1):
- Louisiana State University HSC-Health, School of Dentistry, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Burgess JO, Sadid-Zadeh R, Cakir D, Ramp LC. Clinical evaluation of self-etch and total-etch adhesive systems in noncarious cervical lesions: a two-year report. Oper Dent. 2013 Sep-Oct;38(5):477-87. doi: 10.2341/12-355-CR. Epub 2013 Jan 17. PMID 23327229
- [Background] Lawson NC, Robles A, Fu CC, Lin CP, Sawlani K, Burgess JO. Two-year clinical trial of a universal adhesive in total-etch and self-etch mode in non-carious cervical lesions. J Dent. 2015 Oct;43(10):1229-34. doi: 10.1016/j.jdent.2015.07.009. Epub 2015 Jul 29. PMID 26231300